CLINICAL TRIAL: NCT07405333
Title: Effect of Coughing Exercises Versus Incentive Spirometry on Respiratory Outcomes and Postoperative Recovery Among Children Undergoing Cardiac Surgery.
Brief Title: Effect of Coughing Exercises Versus Incentive Spirometry on Respiratory Function and Recovery in Children After Cardiac Surgery.
Acronym: CEXIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Rusul Khalid Kadim, Graduate Student / Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UOB-NUR-2026-01
Record Dates: First submitted 2026-01-22; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Congenital Heart Disease (CHD); Postoperative Respiratory Dysfunction; Postoperative Recovery After Cardiac Surgery
Keywords: Coughing Exercises; Incentive Spirometry; Congenital Heart Disease; Respiratory Function; Recovery; cardiac surgery; pediatric
MeSH Terms: conditions — Heart Defects, Congenital; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: this is a parallel-assignment randomized interventional study with three arms: coughing exercises, incentive spirometry, and standard care. Participants will remain in their assigned group throughout the study period, receiving the allocated intervention along with standard postoperative care
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coughing Exercises (Experimental): participants in this arm will receive structured postoperative coughing exercises under professional supervision. The exercises include deep breathing followed by effective coughing techniques to enhance airway clearance, promote lung expansion, and prevent postoperative pulmonary complications. The intervention will be performed every 3 hours for three days after cardiac surgery in addition to standard postoperative care.
  Interventions: Behavioral: Coughing Exercises
- Incentive Spirometry (IS) (Experimental): Participants in this arm will receive postoperative incentive spirometry under professional supervision. Children will be instructed to perform slow, deep inhalations using an incentive spirometer to promote lung expansion, improve ventilation. The intervention will be performed 15 times every 3 hours for three days after cardiac surgery in addition to standard postoperative care.
  Interventions: Device: Incentive Spirometry
- Standard Postoperative Care (Active Comparator): Participants in this arm will receive standard postoperative care following cardiac surgery without additional structured respiratory physiotherapy interventions. Standard care includes routine medical and nursing management according to hospital protocols, such as oxygen therapy, pain management, monitoring of vital signs, and general postoperative mobilization as tolerated.
  Interventions: Other: Standard Postoperative Care

INTERVENTIONS:
Behavioral: Coughing Exercises — participants will receive structured postoperative coughing exercises supervised by trained healthcare professionals. The intervention includes instruction on effective deep breathing followed by directed coughing to enhance airway clearance and prevent secretion retention. Exercises will be performed every 3 hours for three consecutive days after cardiac surgery, in addition to standard postoperative care.
  Arms: Coughing Exercises
Device: Incentive Spirometry — participants will perform postoperative incentive spirometry using a standard incentive spirometer under professional supervision. Children will be instructed to perform slow, deep inspirations with visual feedback to promote lung expansion and alveolar recruitment. The intervention will be conducted 15 times every 3 hours for three days after surgery, alongside standard postoperative care.
  Arms: Incentive Spirometry (IS)
Other: Standard Postoperative Care — Participants will receive routine postoperative care according to institutional protocols following cardiac surgery. This includes standard medical and nursing management such as oxygen therapy, pain control, monitoring of vital signs, and mobilization as tolerated, without additional structured respiratory physiotherapy interventions.
  Arms: Standard Postoperative Care

SUMMARY:
This study examines the effects of coughing exercises and incentive spirometry (IS) on lung function and recovery in children who undergo heart surgery. The main goals are to see:

How coughing exercises and IS affect breathing and lung function after surgery? How these exercises influence overall recovery after surgery? Children who participate will be randomly assigned to one of three groups: coughing exercises, IS, or standard care. Those in the exercise groups will perform their assigned breathing exercises every 3 hours for the first 3 days after surgery. Daily check-ups will be conducted to monitor their progress, lung function, and oxygen levels.

The study will measure breathing ability, oxygen levels, and recovery milestones to find out which method is most effective in preventing lung complications and helping children recover faster.

DETAILED DESCRIPTION:
This clinical trial evaluates the effects of coughing exercises and incentive spirometry (IS) on postoperative respiratory outcomes and recovery in children undergoing elective cardiac surgery with cardiopulmonary bypass.

The study aims to answer:

How do coughing exercises and IS influence lung function and breathing after surgery? How do they affect overall recovery, including physical comfort, oxygenation, and prevention of pulmonary complications?

Eligible children aged 6 to 18 years will be randomly assigned to one of three groups:

Coughing exercises group Incentive spirometry group Standard care group Children in the intervention groups will perform the assigned exercises every 3 hours for the first 3 days after surgery. All participants will receive daily monitoring, including vital signs, oxygen saturation, lung function assessment, and observation of postoperative recovery indicators such as feeding tolerance and mobility.

The study will assess primary outcomes such as postoperative respiratory function using a standardized respiratory score, and secondary outcomes including postoperative recovery indicators (quality of recovery scores), incidence of pulmonary complications, and length of stay in the pediatric intensive care unit (ICU).

This research will help identify the most effective method for improving respiratory outcomes, reducing complications, and supporting faster recovery in children after cardiac surgery.

ELIGIBILITY:
Inclusion Crit

* Children aged 6 to 18 years scheduled for elective cardiac surgery.
* Postoperative extubation within 24 hours and judged clinically stable to begin respiratory therapy.
* Hemodynamically stable.

Exclusion Criteria:

* Pre-existing moderate-to-severe chronic lung disease requiring baseline oxygen therapy.
* Neuromuscular disorders significantly impairing cough/inspiratory effort.
* Emergency surgery, ongoing major bleeding.
* Prolonged mechanical ventilation >72 hours or tracheostomy on admission.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-12-07 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Respiratory Function Score. | Baseline, 1 hour after intervention, 3 hours, 6 hours, 24 hours, 48 hours, and 72 hours.
  A composite postoperative respiratory function score assessed using standardized pediatric respiratory severity score, including respiratory rate (breaths/min), oxygen saturation measured by pulse oximetry (SpO₂, %), presence of wheezing (yes/no), use of accessory respiratory muscles (yes/no), and feeding tolerance. Higher scores indicate better respiratory function.

SECONDARY OUTCOMES:
Postoperative Recovery Indicators Assessed by Clinical and Functional Parameters | Baseline, postoperative day 1, and postoperative day 7
  Postoperative quality of recovery assessed using the Pediatric Quality of Recovery (PQoR) scale, which evaluates postoperative pain, comfort, emotional status, physical activity, and feeding tolerance through age-appropriate assessment and caregiver reporting. Higher scores indicate better postoperative recovery.
Length of Intensive Care Unit (ICU) Stay | From ICU admission after surgery until ICU discharge, up to postoperative day 14
  The duration of stay in the pediatric intensive care unit following cardiac surgery, calculated in days from ICU admission to ICU discharge based on hospital medical records..

CONTACTS AND LOCATIONS:
Locations (4):
- Iraq (4):
  - Ibn Al-Bitar Specialized Hospital for Cardiac Surgery, Baghdad, Baghdad Governorate
  - Ibn Al-Nafis Hospital for Cardiac, Thoracic and Vascular Surgery, Baghdad, Baghdad Governorate
  - Iraqi Center for Heart Diseases, Baghdad, Baghdad Governorate
  - Imam Al-Hassan Al-Mujtaba Hospital, Karbala, Karbala Governorate

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of pediatric health information and to protect participant confidentiality. The study involves children undergoing cardiac surgery, and sharing detailed clinical data could risk identification of participants despite de-identification measures. Additionally, no institutional approval has been obtained for secondary use of these data..